CLINICAL TRIAL: NCT05013450
Title: A Phase 1b/2 Trial of Dupilumab Given in Conjunction With PD-1 or PD-L1 Blockade and Anakinra in the Treatment of Relapsed/Refractory Metastatic NSCLC
Brief Title: Dupilumab_Metastatic NSCLC
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Thomas Marron (Other)
Responsible Party: Sponsor-Investigator, Thomas Marron, Director, Early Phase Trials Unit, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-21-00907
Record Dates: First submitted 2021-08-13; First posted 2021-08-19 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — dupilumab; Immune Checkpoint Inhibitors; Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dupilumab + anti-PD-1/PD-L1 (SOC) (Experimental): Patients will continue SOC immunotherapy with PD-1/PD-L1 blockade following progression of disease, and three q3w cycles of dupilumab will be administered
  Interventions: Drug: Dupilumab; Drug: PD-1/PD-L1 blockade
- Anakinra + Dupilumab + anti-PD-1/PD-L1 (SOC) (Experimental): Patients will continue SOC immunotherapy with PD-1/PD-L1 blockade following progression of disease, and three q3w cycles of dupilumab and anakinra will be administered
  Interventions: Drug: Dupilumab; Drug: PD-1/PD-L1 blockade; Drug: Anakinra

INTERVENTIONS:
Drug: Dupilumab — three q3w cycles
Drug: PD-1/PD-L1 blockade — SOC immunotherapy with PD-1/PD-L1 blockade
Drug: Anakinra — 100 mg daily injection for Three q3w cycles
  Arms: Anakinra + Dupilumab + anti-PD-1/PD-L1 (SOC)

SUMMARY:
This is a multi cohort, sequential enrollment clinical trial to determine the safety and tolerability of Dupilumab and Anakinra with PD-(L)1 blockade for patients with relapsed/refractory metastatic NSCLC. For Phase 2, to determine the effect of adding IL-4Ra and IL-1R blockade to PD-(L)1 blocking agents in patients with relapsed/refractory NSCLC, who have progressed on prior PD-(L)1 agents.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a pathologically confirmed diagnosis of NSCLC
* Patients must have progressed (clinically or radiographically) on or following prior therapy with a PD-1 or PD-L1 targeted antibody
* Patients may have only 0 or 1 intervening lines of therapy from the prior PD-(L)1 blocking therapy
* Patient must be willing and able to provide blood samples (12 green-top tubes, roughly 100mL) at the time points indicated in the Study Calendar.
* Patient must be willing and able to have core needle biopsies, or forceps biopsies if clinically feasible by (Goal 3-6 biopsies, final number to be determined by the interventionalist performing the procedure as safe) of tumor prior to initiation of dupilumab and at the on-treatment time point. Should patients undergo pre-treatment or on-treatment biopsy procedure, and inadequate number of biopsies are obtained, they may proceed with initiation/continuation of treatment at the discretion of the investigator and treating physician
* Age ≥ 18 years.
* ECOG 0-2. The exception will be patients carrying long term disability (such as cerebral palsy) where the disability is not acute nor progressive, and unlikely to significantly affect their response to therapy.
* Women of child-bearing potential and men must agree to use adequate contraception prior to study entry, for the duration of study participation, and for 3 months following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:
* Has not undergone a hysterectomy or bilateral oophorectomy; or
* Has not been naturally postmenopausal for at least 12 consecutive months
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Patients who have had chemotherapy within 14 days from start of therapy.
* Palliative radiotherapy is permitted at any time, if deemed in the best interest of the patient.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring antibiotics (exception is a brief (≤10days) course of antibiotics to be completed before initiation of treatment), symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. Patients on chronic steroids (more than 4 weeks at stable dose) equivalent to ≤ 10mg prednisone will not be excluded.
* Has active autoimmune disease that has required systemic treatment in the past 1 year (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is acceptable.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator.
* HIV positive with detectable viral load, or anyone not on stable anti-viral (HAART) regimen, or with <350 CD4+ T cells/microliter in the peripheral blood. HIV testing is not required for patients with no known history of HIV.
* Has known active Hepatitis B (e.g., HBV detected by PCR or active Hepatitis C (e.g., HCV RNA [qualitative] is detected). Patients with hepatitis B (HepBsAg+) who have controlled infection (serum hepatitis B virus DNA PCR that is below the limit of detection AND receiving anti-viral therapy for hepatitis B) are permitted. Patients with controlled infections must undergo periodic monitoring of HBV DNA. Patients must remain on anti-viral therapy for at least 6 months beyond the last dose of investigational study drug.
* History of allogeneic hematopoietic cell transplantation or solid organ transplantation.
* Receipt of a live vaccine within 30 days of planned start of study medication
* Documented allergic or hypersensitivity response to any protein therapeutics (e.g., recombinant proteins, vaccines, intravenous immune globulins, monoclonal antibodies, receptor traps)Principle investigator believes that for one or multiple reasons the patient will be unable to comply with all study visits, or if they believe the trial is not clinically in the best interest of the patient.
* History of irAE in response to prior immunotherapy that has not improved to a Grade 0 or 1; this does not include chronic conditions such as endocrinopathies which can be treated with hormone replacement therapy
* History of interstitial lung disease (e.g., idiopathic pulmonary fibrosis, organizing pneumonia) or active, noninfectious pneumonitis attributed to prior use of cancer immunotherapy that required immune-suppressive doses of glucocorticoids to assist with management. A history of radiation pneumonitis in the radiation field is permitted.
* Patient has received Anakinra in the last 12 months (Cohort B).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2025-09-10 (Actual); Study Completion 2025-12-09 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLTs) | 9 weeks
  Phase 1: Dose Limiting Toxicity (DLTs) as defined based on the NCI Common Toxicity Criteria for Adverse Events (CTCAE), version 5.0.
Overall Response Rate (ORR) | 9 weeks
  Phase 2: Overall response rate by imaging at time of first repeat imaging (~9w from the start of therapy) using standard response criteria (RECIST v1.126). ORR is defined as the combined percent of the patients experiencing a partial response (PR) or a complete response (CR) at time of first reimaging.

SECONDARY OUTCOMES:
Best overall response (BORR) | 2 years
  Best overall response (BORR) will be a combined percent of the patients experiencing a partial response (PR) or a complete response (CR) at any point within the first year from the initiation of therapy, or until the documented progression of disease or start of a new anti-cancer therapy.
Progression-free survival (PFS) | 2 years
  Progression-free survival (PFS) is defined as the time in days from the first administration of dupilumab until documented progression of disease on imaging or death Defined as the time in days from the first administration of dupilumab until documented progression of disease on imaging or death
Overall Survival (OS) | 2 years
  Overall survival (OS) is defined as the time in days from the first administration of dupilumab until documented death from any cause.
Duration of response (DOR) | 2 years
  Duration of response (DOR) is defined as the time from which a patient achieves either a PR or a CR until subsequent progression of disease is documented radiographically or clinically.
  Defined as the time from which a patient achieves either a PR or a CR until subsequent progression of disease is documented radiographically or clinically.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Marron, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Tisch Cancer Institute, Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ('learned intermediary') identified for this purpose. For individual participant data meta-analysis. Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata. Information regarding submitting proposals and accessing data may be found at (Link to be included in the URL field below).

REFERENCES:
- [Derived] LaMarche NM, Hegde S, Park MD, Maier BB, Troncoso L, Le Berichel J, Hamon P, Belabed M, Mattiuz R, Hennequin C, Chin T, Reid AM, Reyes-Torres I, Nemeth E, Zhang R, Olson OC, Doroshow DB, Rohs NC, Gomez JE, Veluswamy R, Hall N, Venturini N, Ginhoux F, Liu Z, Buckup M, Figueiredo I, Roudko V, Miyake K, Karasuyama H, Gonzalez-Kozlova E, Gnjatic S, Passegue E, Kim-Schulze S, Brown BD, Hirsch FR, Kim BS, Marron TU, Merad M. An IL-4 signalling axis in bone marrow drives pro-tumorigenic myelopoiesis. Nature. 2024 Jan;625(7993):166-174. doi: 10.1038/s41586-023-06797-9. Epub 2023 Dec 6. PMID 38057662

DOCUMENTS (1):
  • Informed Consent Form (2025-07-08): https://cdn.clinicaltrials.gov/large-docs/50/NCT05013450/ICF_000.pdf